CLINICAL TRIAL: NCT05680636
Title: A New Clinical Score for Deep Vein Thrombosis: the Role of Differential Leg Skin Temperature Measured With Handheld Low-cost Infrared Thermometers.
Brief Title: New Clinical Score for Deep Vein Thrombosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Accademia Italiana Medicina Osteopatica (Other)
Responsible Party: Principal Investigator, ALESSANDRA ABENAVOLI, Head of Research, Accademia Italiana Medicina Osteopatica
Other Study IDs: 002
Record Dates: First submitted 2022-09-21; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: temperature measurement — Differential Leg Skin Temperature Measured With Handheld Low-cost Infrared Thermometers.

SUMMARY:
A new Clinical Score (CS) to rule out Deep Vein Thrombosis (DVT) has to be derived and internally validated (with bootstrap method), from patients suspected of DVT in Italy. Primary care physicians (general practitioners) in Lombardy will be instructed to inform patients suspected of DVT about this research and get in touch with the team to get details and, eventually, volunteer for the study. The CS includes categorical variables and a continuous variable: the differential leg skin temperature measured with a low-cost handheld infrared thermometer in object surface mode.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected of deep vein thrombosis.

Exclusion Criteria:

* under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Suspicion of deep vein thrombosis should be based on the presence of at least one of the following signs/symptoms
  * unilateral swelling of the lower limbs
  * unilateral erythema of the lower limbs
  * unilateral pain in the lower limbs
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01-21 (Estimated); Primary Completion 2023-09-21 (Estimated); Study Completion 2023-09-21 (Estimated)

PRIMARY OUTCOMES:
presence of DVT | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Mapelli, Bsc (HOns), Principal Investigator — Accademia Italiana Medicina Osteopatica
Locations (1):
- Studio Medico, Gessate, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided